CLINICAL TRIAL: NCT01791660
Title: Targeted Fat Reduction of Pseudogynecomastia in the Male Breast Using the ZELTIQ Coolsculpting System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dermatology, Laser & Vein Specialists of the Carolinas (Other)
Responsible Party: Principal Investigator, Girish Munavalli, MD MHS, MD,MHS, Dermatology, Laser & Vein Specialists of the Carolinas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLVSC-ZA-001
Record Dates: First submitted 2012-08-31; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Gynecomastia
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zeltiq Coolsculpting System (Experimental): non-invasive device designed to cool subcutaneous fat without affecting adjacent or underlying structures.
  Interventions: Device: Zeltiq Coolsculpting System

INTERVENTIONS:
Device: Zeltiq Coolsculpting System — Non-invasive device designed to cool subcutaneous fat without affecting adjacent or underlying structures.

SUMMARY:
Protocol is intended for the clinical evaluation of fat reduction in male breasts (pseudogynecomastia) using the ZELTIQ Coolsculpting System. The ZELTIQ Coolsculpting system has received market clearance from the U.S.FDA for non-invasive fat layer reduction in the flanks, and is commercially available.

Primary study endpoint is changes in the shape and reduction of the fat in the breast as established by photographic imaging and ultrasound imaging of the treated area.

Secondary endpoints will provide supportive data to evaluate device performance (subject satisfaction & fat reduction measured with ultrasound).

DETAILED DESCRIPTION:
not desired

ELIGIBILITY:
Inclusion Criteria:

* INCLUDED:

  1. Male subjects > 18 years of age and < 70 years of age.
  2. Subject has clearly visible, palpable, excess fatty tissue in their breast area, and minimal fibrous tissue.
  3. Subject has not had weight change exceeding 10 pounds in the preceding month.
  4. Subject agrees to maintain their weight (i.e., within +/- 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
  5. Subject has read and signed a written informed consent form.

     Exclusion Criteria:

     EXCLUDED:

  <!-- -->

  1. Subject has had a surgical procedure(s) in the area of intended treatment.
  2. Subject has had an invasive fat reduction procedure (e.g., liposuction or mesotherapy) in the area of intended treatment.
  3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment.
  4. Subject needs to administer, or has a known history of, subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
  5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
  6. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
  7. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
  8. Subject body mass index (BMI) exceeds 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
  9. Subject is taking or has taken diet pills or diet supplements within the past month.
  10. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation.
  11. Subject is unable or unwilling to comply with the study requirements.
  12. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
  13. Personal history of previous breast malignancy.
  14. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.
  15. Subject is taking any medication which could cause abnormal breast enlargement - including but not limited to: digoxin, furosemide, gonadotropins, clomiphene, phenytoin, and exogenous testosterone, ketoconazole, metronidazole, alkylating agents, cisplatin, spironolactone, cimetidine, flutamide, finasteride, etomidate, isonicotinic acid hydrazide, methyldopa, busulfan, tricyclic antidepressants, diazepam, penicillamine, omeprazole, phenothiazines, calcium channel blockers, angiotensin-converting enzyme (ACE) inhibitors.
  16. Recent history (within the past 5 years) of substance abuse (alcohol, marijuana or heroin).
  17. Subject has no history of the following medical conditions: Klinefelter syndrome, Congenital anorchia, Testicular trauma, Testicular torsion, Viral orchitis, Kallmann syndrome , Pituitary tumors, Malignancies that increase the serum level of hCG (eg, large cell lung cancer, gastric carcinoma, renal cell carcinoma, hepatoma), Renal failure, Hyperthyroidism, Malnutrition, Androgen insensitivity syndrome, Five-alpha-reductase deficiency syndrome

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
reduction of the fat layer | 8 months
  Visual, photographic and ultrasound measured changes in the shape and reduction of the fat in the male breast.

SECONDARY OUTCOMES:
visual reduction of the fat layer | 8 months
  Subject satisfaction measured by subject questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Girish S Munavalli, MD MHS, Principal Investigator — Dermatology, Laser & Vein Specialists of the Carolinas
Locations (1):
- Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina, United States

REFERENCES:
- See also: related information — http://www.carolinaskin.com